CLINICAL TRIAL: NCT07011342
Title: Utility of 18F-rhPSMA-7.3 in the Diagnosis of Prostate Cancer After Focal Gland Treatment
Acronym: SCOUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Blue Earth Diagnositcs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCOUT-IIT; Pro2024-0305 (Other: HMH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-rhPSMA-7.3 (Experimental): Patients will undergo a PSMA-PET scan at 1 year (+/- 60 days) after treatment with SOC focal therapy using a radiohybrid Prostate-Specific Membrane Antigen (rhPSMA)-targeted PET scan using 18F-rhPSMA-7.3 (Posluma).
  The rhPSMA-targeted PET scan is an FDA-approved PET scan to detect the presence of lesions positive for prostate-specific membrane antigen (PSMA) in men with prostate cancer. 18F-rhPSMA-7.3 (Posluma) injection is a radioactive diagnostic agent that is administered in the form of an intravenous injection.
  Interventions: Drug: 18F-rhPSMA-7.3

INTERVENTIONS:
Drug: 18F-rhPSMA-7.3 — Utility of 18F-rhPSMA-7.3 in the diagnosis of prostate cancer after Focal Gland Treatment (SCOUT)

SUMMARY:
To evaluate the effectiveness of a PSMA-PET scan in identifying recurrent prostate cancer after focal therapy

DETAILED DESCRIPTION:
PSMA is a protein that is highly expressed in prostate cancer cells, making it an excellent specific target for imaging with PET scans that can provide detailed information about the location, extent and aggressiveness of prostate cancer lesions. These scans have proven invaluable for identifying and characterizing prostate cancer, aiding in treatment planning, and Monitoring treatment response. It's true and fully utility in focal therapy for prostate cancer is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years or older;
* Patient must have a pre-treatment MRI;
* Patient underwent SOC focal therapy with either focal or hemiablation for the treatment of intermediate risk prostate cancer in the past 9 months prior to enrollment;
* Intermediate risk disease as defined by American Urology Academy (AUA)/National Comprehensive Cancer Network (NCCN) guidelines (see Appendix A)
* Life Expectancy of 10 years or more;
* Underwent standard template biopsy before treatment with a minimum of 2 cores into the MRI visible lesion if lesion was present;
* Patient understands the purpose of the trial and procedures required for the trial, and can provide signed informed consent as which includes compliances with the requirements and restrictions listed in the informed consent form (ICF) and in the study protocol; and
* Ability to adhere to the study visit schedule and all the protocol requirements, including surveillance imaging and test specimen (blood sample) collection at specified time points.

Exclusion Criteria:

* Patients under the age of 18 will be considered pediatric patients and will not be included in this study because they are thought to represent a unique population outside the scope of this study as it is aimed at identifying factors that affect adults only.
* Patients previously treated with whole gland ablation or prior partial gland ablation over 9 months prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of PSMA-PET scan in identifying recurrent prostate cancer after focal therapy | Approximately 1 year after SOC focal therapy.
  All patients will get a biopsy to assess the effectiveness of treatment at 1 year, which is standard protocol at our institutions (all patients undergo biopsy at year 1 and 3 at our institutions). The post-treatment PSMA-PET scan will be correlated to 1-year biopsy results to study the utility of such a scan. Recurrence is defined by a positive PSMA-PET scan and positive biopsy in the area of PET scan tracer uptake at 1 year after SOC focal treatment.

SECONDARY OUTCOMES:
To report the sensitivity and specificity in evaluating PSMA-PET scan | Approximately 1 year after SOC focal therapy.
  Sensitivity and specificity will be reported under the ROC and AUC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Yerrman, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Hopstaken JS, Bomers JGR, Sedelaar MJP, Valerio M, Futterer JJ, Rovers MM. An Updated Systematic Review on Focal Therapy in Localized Prostate Cancer: What Has Changed over the Past 5 Years? Eur Urol. 2022 Jan;81(1):5-33. doi: 10.1016/j.eururo.2021.08.005. Epub 2021 Sep 4. PMID 34489140
- [Background] Nguyen-Nielsen M, Borre M. Diagnostic and Therapeutic Strategies for Prostate Cancer. Semin Nucl Med. 2016 Nov;46(6):484-490. doi: 10.1053/j.semnuclmed.2016.07.002. Epub 2016 Sep 3. PMID 27825428
- [Background] Chang SS. Overview of prostate-specific membrane antigen. Rev Urol. 2004;6 Suppl 10(Suppl 10):S13-8. PMID 16985927
- [Background] Cereser L, Evangelista L, Giannarini G, Girometti R. Prostate MRI and PSMA-PET in the Primary Diagnosis of Prostate Cancer. Diagnostics (Basel). 2023 Aug 17;13(16):2697. doi: 10.3390/diagnostics13162697. PMID 37627956
- [Background] Kwon DH, Velazquez AI, de Kouchkovsky I. PSMA PET Scan. JAMA Oncol. 2022 Dec 1;8(12):1860. doi: 10.1001/jamaoncol.2022.3531. PMID 36201182
- [Background] Testa U, Castelli G, Pelosi E. Cellular and Molecular Mechanisms Underlying Prostate Cancer Development: Therapeutic Implications. Medicines (Basel). 2019 Jul 30;6(3):82. doi: 10.3390/medicines6030082. PMID 31366128
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Heidenreich A, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Mottet N, Schmid HP, van der Kwast T, Wiegel T, Zattoni F; European Association of Urology. EAU guidelines on prostate cancer. Part 1: screening, diagnosis, and treatment of clinically localised disease. Eur Urol. 2011 Jan;59(1):61-71. doi: 10.1016/j.eururo.2010.10.039. Epub 2010 Oct 28. PMID 21056534
- [Background] Izawa JI, Klotz L, Siemens DR, Kassouf W, So A, Jordan J, Chetner M, Iansavichene AE. Prostate cancer screening: Canadian guidelines 2011. Can Urol Assoc J. 2011 Aug;5(4):235-40. doi: 10.5489/cuaj.11134. No abstract available. PMID 21801679
- [Background] Olleik G, Kassouf W, Aprikian A, Hu J, Vanhuyse M, Cury F, Peacock S, Bonnevier E, Palenius E, Dragomir A. Evaluation of New Tests and Interventions for Prostate Cancer Management: A Systematic Review. J Natl Compr Canc Netw. 2018 Nov;16(11):1340-1351. doi: 10.6004/jnccn.2018.7055. PMID 30442734
- [Background] Atluri S, Mouzannar A, Venkatramani V, Parekh DJ, Nahar B. Focal therapy for localized prostate cancer - Current status. Indian J Urol. 2022 Jan-Mar;38(1):7-14. doi: 10.4103/iju.iju_166_21. Epub 2022 Jan 1. PMID 35136289
- [Background] Borley N, Feneley MR. Prostate cancer: diagnosis and staging. Asian J Androl. 2009 Jan;11(1):74-80. doi: 10.1038/aja.2008.19. Epub 2008 Dec 1. PMID 19050692
- [Background] Ortner G, Tzanaki E, Rai BP, Nagele U, Tokas T. Transperineal prostate biopsy: The modern gold standard to prostate cancer diagnosis. Turk J Urol. 2021 Feb;47(Supp. 1):S19-S26. doi: 10.5152/tud.2020.20358. Epub 2020 Oct 9. PMID 33052837
- [Background] Moreira LF, Mussi TC, Cunha MLD, Filippi RZ, Baroni RH. Accuracy of 68Ga-PSMA PET/CT for lymph node and bone primary staging in prostate cancer. Urol Oncol. 2022 Mar;40(3):104.e17-104.e21. doi: 10.1016/j.urolonc.2021.11.007. Epub 2021 Dec 13. PMID 34911650
- [Background] Hoffman A, Amiel GE. The Impact of PSMA PET/CT on Modern Prostate Cancer Management and Decision Making-The Urological Perspective. Cancers (Basel). 2023 Jun 29;15(13):3402. doi: 10.3390/cancers15133402. PMID 37444512
- [Background] Lu, Grace,
- [Background] Hanley JA, McNeil BJ. The meaning and use of the area under a receiver operating characteristic (ROC) curve. Radiology. 1982 Apr;143(1):29-36. doi: 10.1148/radiology.143.1.7063747.
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Background] Eastham JA, Auffenberg GB, Barocas DA, Chou R, Crispino T, Davis JW, Eggener S, Horwitz EM, Kane CJ, Kirkby E, Lin DW, McBride SM, Morgans AK, Pierorazio PM, Rodrigues G, Wong WW, Boorjian SA. Clinically Localized Prostate Cancer: AUA/ASTRO Guideline, Part I: Introduction, Risk Assessment, Staging, and Risk-Based Management. J Urol. 2022 Jul;208(1):10-18. doi: 10.1097/JU.0000000000002757. Epub 2022 May 10. PMID 35536144
- [Background] National Comprehensive Cancer Network. Prostate Cancer (Version 4.2024). May 17, 2024]; Available from: https://www.nccn.org/professionals/physician_gls/pdf/prostate.pdf.